CLINICAL TRIAL: NCT02263092
Title: Effects of Transcranial Direct Current Stimulation Associated With Physical Exercise: a Metaplasticity Study
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Kátia Monte-Silva, PHD, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: Exercise_tdcs_metaplasticity
Record Dates: First submitted 2014-08-30; First posted 2014-10-13 (Estimated); Last update posted 2015-02-26 (Estimated); Status verified 2014-05

CONDITIONS: Metaplasticity; Healthy Subjects
Keywords: Cortical excitability; Plasticity; Healthy subjects
MeSH Terms: interventions — Exercise; Transcranial Direct Current Stimulation; RE1-silencing transcription factor

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (10):
- 15 minutes of physical exercise (Experimental): the subjects will do physical exercise on a treadmill with 64 to 74% of maxHR
  Interventions: Behavioral: Physical exercise
- 10 minutes of physical exercise (Experimental): - the subjects will do physical exercise on a treadmill with 77 to 95% of maxHR.
  Interventions: Behavioral: Physical exercise
- 30 minutes of physical exercise (Experimental): - the subjects will do physical exercise on a treadmill with 57 to 63% of maxHR.
  Interventions: Behavioral: Physical exercise
- Rest/control (Experimental): the subjects will be on 15 or 30 minutes seat without move the legs.
  Interventions: Behavioral: Rest
- Anodal tDCS + physical exercise 1 (Experimental): the subjects will be undergo to anodal tDCS + physical exercise 1
  Interventions: Behavioral: Physical exercise; Device: tDCS
- Anodal tDCS + physical exercise 2 (Experimental): the subjects will be undergo to anodal tDCS + physical exercise 2
  Interventions: Behavioral: Physical exercise; Device: tDCS
- Cathodal tDCS + physical exercise 1 (Experimental): the subjects will be undergo to cathodal tDCS + physical exercise 1
  Interventions: Behavioral: Physical exercise; Device: tDCS
- Cathodal tDCS + physical exercise 2 (Experimental): - the subjects will be undergo to cathodal tDCS + physical exercise 2
  Interventions: Behavioral: Physical exercise; Device: tDCS
- Sham tDCS + physical exercise 1 (Experimental): the subjects will be undergo to sham tDCS + physical exercise 1
  Interventions: Behavioral: Physical exercise; Device: tDCS
- Sham tDCS + physical exercise 2 (Experimental): the subjects will be undergo to sham tDCS + physical exercise 2
  Interventions: Behavioral: Physical exercise; Device: tDCS

INTERVENTIONS:
Behavioral: Physical exercise — The intensity of physical exercise will be determine by the maximum heart rate (max HR) using the formula (220 - age). For the high intensity, the intensity will between 79-95% xx% of maxHR; moderate intensity, 64-76% of maxHR; mild intensity, 57-63% of maxHR. Furthermore, during the physical exercise the heart rate will be continuous evaluate by the POLAR and the rate perceived scale will be register in each 3 minutes by the modified Borg scale
  Arms: 10 minutes of physical exercise; 15 minutes of physical exercise; 30 minutes of physical exercise; Anodal tDCS + physical exercise 1; Anodal tDCS + physical exercise 2; Cathodal tDCS + physical exercise 1; Cathodal tDCS + physical exercise 2; Sham tDCS + physical exercise 1; Sham tDCS + physical exercise 2
Device: tDCS — Current will be applied by a DC stimulator (NeuroConn, Germany) using a pair of saline-soaked sponge electrodes (surface 35 and 36cm²). tDCS will be applied to Cz and Oz according to International 10-20 EEG system. In the anodal tDCS, the anode will be placed in Cz and cathode in Oz. In the cathodal tDCS the inverse position will be done. Parameters of current intensity and duration (dose) used were 2 mA stimulation intensity for 20 minutes with current ramping up and down of 10 seconds each.For sham, the same position of anodal tDCS will be assumed, however, current duration is only 30 seconds, with current ramping up and down of 10 seconds each. Moreover, the electrostimulation device is automatically turned off without patient's perception. Thus, patients experience early sensations (mild to moderate tingling) in stimulation site without inducing effect. Moreover, after each tDCS session, patients will answer adverse effects questionnaire.
  Arms: Anodal tDCS + physical exercise 1; Anodal tDCS + physical exercise 2; Cathodal tDCS + physical exercise 1; Cathodal tDCS + physical exercise 2; Sham tDCS + physical exercise 1; Sham tDCS + physical exercise 2
Behavioral: Rest — 15 or 30 minutes seat without move the legs
  Arms: Rest/control

SUMMARY:
This study aims to understand metaplasticity through the association of transcranial direct current stimulation (tDCS) and physical exercise. For this purpose, the study will be separate in 2 phases: in the first phase the aim is verify the effects of physical exercise on cortical excitability. After this 1st phase two intensities of physical exercise will be chosen for the second phase. In the 2nd phase, subjects will undergo to anodal, cathodal and sham tDCS plus physical exercise.

DETAILED DESCRIPTION:
Before the two phases of the study, the subjects will be evaluate in the following aspects: anxiety by the beck anxiety inventory; depression by the beck depression inventory; level of physical exercise by the international physical activity questionnaire; stress by the stress perceived scale 10.

In the first phase, the subjects will be undergo to 4 conditions: (i) 15 minutes of physical exercise with moderate intensity; (ii) 10 minutes of physical exercise with high intensity; (iii) 30 minutes of physical exercise with mild intensity; (iv) 15 or 30 minutes of rest. Before each condition, cortical excitability will be measure through the Transcranial magnetic stimulation by motor evoked potential (MEP); the blood glucose level will be evaluate by glucometer. The MEP also will be done immediately after the physical exercise and in every 5 min for 30 after the end of exercise/rest. The blood glucose level will be done immediately after the exercise..

In the second phase, the subjects will be undergo to 6 conditions: (i) anodal tDCS + physical exercise 1; (ii) anodal tDCS + physical exercise 2; (iii) cathodal tDCS + physical exercise 1; (iv) cathodal tDCS + physical exercise 2; (v) sham tDCS + physical exercise 1; (vi) sham tDCS + physical exercise 2. The intensity and time of physical exercise depends of the results of the previous phase and will be determine after the end of phase 1. In this phase, the blood glucose level will be evaluate before and immediately the physical exercise. The cortical excitability will be evaluate through the Transcranial magnetic stimulation by the following measures: motor evoked potential - before the tDCS,after tDCS, immediately , 10, 20, 30, 60, 90 minutes after the exercise; resting motor threshold - before tdcs, immediately and 90 minutes after the exercise; recruitment curve - before tdcs, immediately and 90 minutes after the exercise.

tDCS condition During tDCS application, patients will be seated in a comfortable chair with head and arms rests. Current will be applied by a DC stimulator (NeuroConn, Germany) using a pair of saline-soaked sponge electrodes (surface 35 and 36cm²).

tDCS will be applied to Cz and Oz according to International 10-20 EEG system. In the anodal tDCS, the anode will be placed in Cz and cathode in Oz. In the cathodal tDCS the inverse position will be done. Parameters of current intensity and duration (dose) used were previously established in poststroke patients: 2 mA stimulation intensity for 20 minutes with current ramping up and down of 10 seconds each.

Sham tDCS has been used in several studies to evaluate the effect of active tDCS. For sham, the same position of anodal tDCS will be assumed, however, current duration is only 30 seconds, with current ramping up and down of 10 seconds each. Moreover, the electrostimulation device is automatically turned off without patient's perception. Thus, patients experience early sensations (mild to moderate tingling) in stimulation site without inducing effect. Moreover, after each tDCS session, patients will answer adverse effects questionnaire.

Physical exercise condition The intensity of physical exercise will be determine by the maximum heart rate (max HR) using the formula (220 - age). For the high intensity, the intensity will between xx and xx% of maxHR; moderate intensity, 64-76% of maxHR; mild intensity, 57-63% of maxHR. Furthermore, during the physical exercise the heart rate will be continuous evaluate by the POLAR and the rate perceived scale will be register in each 3 minutes by the modified Borg scale Outcome measures Evaluation of brain activity will be performed using single-pulse transcranial magnetic stimulation (TMS-p). Magnetic stimulation (Neurosoft, Russia) will be applied through a figure-8 coil to determine motor cortex representation of right tibial anterior muscle (hotspot) and performed the following electrophysiological measures to assess cortical activity: (i) Motor Evoked Potential (MEP); (ii) resting motor threshold (RMT) and (iii) Recruitment curve (RC).

Firstly, patients will be instructed to sit in a chair and to search a comfortable position. The hotspot will be considered the most excitable area, with more intense motor evoked potential (MEP), measured by electromyography.

The following electrophysiological measures will be performed in left cerebral hemisphere to assess cortical activity:

(i) Motor Evoked Potential (MEP) : the intensity of magnetic stimulator is adjusted to produce an average MEP of 0.4 mV. TMS-p will be applied in the area of cortical representation of the tibial anterior and mean responses to stimuli should reach 0.4 to 0.6 mV.

(ii) Resting motor threshold (RMT) : will be request to the patient to perform contraction of the tibial anterior muscle and then, will be given ten pulses by TMS-p to determinate resting motor threshold. Motor threshold corresponds to the lowest intensity of TMS-p to produce a MEP of 50μV in 50% of the pulses applied to the hotspot.

(iii) Recruitment curve (RC): Five stimuli were applied at each of the following intensities: 5% below resting motor threshold (RMT), RMT, 5% above RMT, 10% above RMT, 20% above RMT, 30% above RMT, 35% above RMT and at 100% of stimulator output. The five stimuli at each intensity were delivered in a block, but the order of stimulation intensity changes was random. The interval between successive TMS stimuli was between 5.5 to 6.5 s.

ELIGIBILITY:
Inclusion Criteria:

* Self reported healthy
* Right handed

Exclusion Criteria:

* Prior neurological diseases
* Multiple brain lesions
* Metal implant in the skull and face
* Pacemaker
* History of seizures
* Epilepsy
* Pregnancy
* Hemodynamic instability
* Use of medications which change the cortical excitability, such as antidepressants, anxiolytics.
* Energy expenditure > 3000 METS

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2014-02; Primary Completion 2015-02 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Change on cortical excitability - motor evoked potential (MEP) | Phase 1 - in each session (every day), baseline and every 5 minutes for 30 minutes after exercise/rest. Phase 2 - in each session (every day), baseline, after, 10, 20, 30, 60 and 90 after tDCS + exercise

SECONDARY OUTCOMES:
Change on cortical excitability - resting motor threshold (RMT) | Phase 2 - in each session (every day), baseline, after and 90 after tDCS + exercise
Change on cortical excitability - Recruitment curve (RC) | Phase 2 - in each session (every day), baseline, after and 90 after tDCS + exercise

CONTACTS AND LOCATIONS:
Overall Officials: Kátia Monte-Silva, PHD, Study Director — Applied Neuroscience Laboratory, Universidade Federal de Pernambuco
Locations (1):
- Applied Neuroscience Laboratory, Universidade Federal de Pernambuco, Recife, Pernambuco, Brazil